CLINICAL TRIAL: NCT04096716
Title: Mapping Draining Lymph Nodes in CNS Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient funding/staff
Sponsor: Washington University School of Medicine (Other)
Collaborators: Lloyd J. Old STAR Program (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201908018
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Central Nervous System Neoplasms; Central Nervous System Tumor
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1: Tc-99m tilmanocept (Experimental): * The surgeon will inject up to 0.5 mL of reconstituted Tc-99m tilmanocept using a blunt tipped needle 1 cm into the wall of the resection cavity after completing surgical resection of the tumor
  * Portable planar imaging will be obtained at 4.5 ± 2.5 hours and 24 +/- 8 hours after injection of Tc-99m tilmanocept.
  Interventions: Drug: Tc-99m tilmanocept
- Cohort 2A: Tc-99m tilmanocept frontal lobe injection site (Experimental): * The surgeon will inject up to 0.5 mL of reconstituted Tc-99m tilmanocept using a blunt tipped needle 1 cm into the wall of the resection cavity after completing surgical resection of the tumor
  * SPECT/CT of the head and neck will be obtained when practical on the day of surgery.
  If the patient is not sufficiently recovered from surgery to be transported to the Division of Nuclear Medicine for imaging, SPECT/CT will be done on Day 2
  Interventions: Drug: Tc-99m tilmanocept
- Cohort 2B: Tc-99m tilmanocept parietal lobe injection site (Experimental): * The surgeon will inject up to 0.5 mL of reconstituted Tc-99m tilmanocept using a blunt tipped needle 1 cm into the wall of the resection cavity after completing surgical resection of the tumor
  * SPECT/CT of the head and neck will be obtained when practical on the day of surgery.
  If the patient is not sufficiently recovered from surgery to be transported to the Division of Nuclear Medicine for imaging, SPECT/CT will be done on Day 2
  Interventions: Drug: Tc-99m tilmanocept
- Cohort 2C: Tc-99m tilmanocept temporal lobe injection site (Experimental): * The surgeon will inject up to 0.5 mL of reconstituted Tc-99m tilmanocept using a blunt tipped needle 1 cm into the wall of the resection cavity after completing surgical resection of the tumor
  * SPECT/CT of the head and neck will be obtained when practical on the day of surgery.
  If the patient is not sufficiently recovered from surgery to be transported to the Division of Nuclear Medicine for imaging, SPECT/CT will be done on Day 2
  Interventions: Drug: Tc-99m tilmanocept
- Cohort 2D: Tc-99m tilmanocept occipital lobe injection site (Experimental): * The surgeon will inject up to 0.5 mL of reconstituted Tc-99m tilmanocept using a blunt tipped needle 1 cm into the wall of the resection cavity after completing surgical resection of the tumor
  * SPECT/CT of the head and neck will be obtained when practical on the day of surgery.
  If the patient is not sufficiently recovered from surgery to be transported to the Division of Nuclear Medicine for imaging, SPECT/CT will be done on Day 2
  Interventions: Drug: Tc-99m tilmanocept
- Cohort 3: Tc-99m tilmanocept stereotactic needle biopsy of tumor (Experimental): * The surgeon will inject up to 0.3 mL of reconstituted Tc-99m tilmanocept after completing the stereotactic biopsy of the tumor
  * SPECT/CT of the head and neck will be obtained on the day of biopsy, when practical. If the patient is not sufficiently recovered from biopsy to be transported to the Division of Nuclear Medicine for imaging, SPECT/CT will be done on Day 2
  Interventions: Drug: Tc-99m tilmanocept

INTERVENTIONS:
Drug: Tc-99m tilmanocept — Tc-99m tilmanocept is a radioactive diagnostic agent.
  Other Names: Lymphoseek

SUMMARY:
The purpose of this research study is to determine whether the lymph nodes that drain a brain tumor can be detected by imaging after injection of a substance called Tc-99m tilmanocept directly into the brain tissue around the tumor. Tc-99m tilmanocept is a radioactive substance that is used to find lymph nodes by injecting it and then scanning the body with a device that can trace its radioactivity. In this study, the investigators are looking to see how long it takes the Tc-99m tilmanocept to travel from the tumor to the lymph nodes. The investigators will be using it to map lymph nodes as they relate to specific brain areas.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for surgical resection or stereotactic biopsy of suspected brain tumor, including benign tumors (e.g., meningioma) and malignant tumors (e.g., glioma or metastatic disease).
* Suitable candidate to receive Tc-99m tilmanocept injection and study related imaging post-operatively per the Principal Investigator and/or treating neurosurgeon.
* At least 18 years of age.
* Willing and able to provide informed consent (or consent of legally authorized representative).

Exclusion Criteria:

* Documented hypersensitivity to dextran and/or modified forms of dextran.
* Pregnant.
* Prior surgical evacuation of lymph nodes of the head and/or neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Time course of Tc-99m tilmanocept drainage to the lymph nodes from the brain (Cohort 1 only) | Up to Day 2
Identify and map lymph nodes from distinct brain regions as measured by the 2013 international consensus guidelines for cervical and cranial lymph nodes | Up to Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Tanner Johanns, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu